CLINICAL TRIAL: NCT07045025
Title: Prevalence of Endodontic Procedural Errors Using CBCT in an Egyptian Subpopulation: A Cross-Sectional Study
Brief Title: Endodontic Errors Detected by CBCT in Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esbah Adam Ahmed Mohamed, Master Degree Candidate in Endodontics, Cairo University, Cairo University
Other Study IDs: New ENDO 1-1-1 n/code=7 (3/5 G
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Endodontic Procedural Errors in Root Canal Treated Teeth
Keywords: Prevalence of Endodontic Procedural Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Clinical Intervention - Analysis of Previously Acquired CBCT Scans — This study does not involve any clinical or therapeutic intervention. It is solely based on the retrospective analysis of previously acquired CBCT scans from patients who have undergone root canal treatment. No drugs, devices, or procedures are administered or applied to participants as part of this study.

SUMMARY:
This observational cross-sectional study aims to evaluate the prevalence of endodontic procedural errors in root canal-treated teeth among an Egyptian subpopulation using cone-beam computed tomography (CBCT). The study will analyze CBCT scans obtained from radiology centers in Cairo to detect errors such as missed canals, short fillings, perforations, fractured instruments, and other complications. Understanding the frequency and distribution of these errors between the maxillary and mandibular arches may help improve endodontic treatment outcomes and raise awareness of common procedural challenges. The study does not involve any new treatment or drug but will rely on previously taken CBCT images.

DETAILED DESCRIPTION:
The biological and therapeutic goals of Endodontic treatment are to prevent apical lesions or to establish ideal healing conditions by removing bacteria and infection from the root canal system and preventing reinfection. However, endodontic mishaps such as incorrect diagnosis, missed canals, perforations, instrument separation, over- or under-obturation, and vertical root fractures compromise the success of root canal therapy.

The reported success rate of endodontic treatments by general dentists ranges from 60% to 75%. Procedural errors are a significant factor contributing to the suboptimal success rate of endodontic treatments performed by general dentists. Moreover, the global prevalence of periapical lesion is approximately 52% in individuals and 5% in teeth, with higher frequency in teeth with root-filled teeth compered to non-treated teeth.

Procedural errors may be difficult to correct. Certain procedural errors could need endodontic retreatment, apicoectomy, or even tooth extraction. Root canal transportation, apical perforation, strip perforation, access cavity perforation, and instrument fracture are among the commonly occurring procedural errors. The working length of the root canal filling is a critical factor, with fillings short of the apex by 2 mm reducing success rates to 68-77% and overfills beyond the apex yielding around 75% success rates.

Endodontic treatment for molar teeth is more challenging and requires more caution than anterior and premolar teeth, and is associated with a higher rate of procedural errors. The reason for this is their difficulty in accessibility and anatomical complexity. This is reflected in the distribution of errors, were Procedural errors were more frequently observed in mandibular teeth (53.1%) than maxillary teeth (46.9%), with the highest error rate found in the right and left permanent mandibular first molars (20.2% and 14.3%, respectively).

Cone-beam computed tomography (CBCT) it delivers high-quality images and images providing three-dimensional imaging, allowing detailed views of individual teeth from any angle. This makes it an effective tool for diagnosing, planning, and monitoring endodontic treatment. CBCT can detect periapical radiolucency before they would be apparent on conventional radiographs. While traditional radiographs are less expensive and expose patients to lower radiation doses, research has demonstrated that CBCT images are better for diagnosing periapical lesions.

Rationale for conducting the research:

In Egypt, there is a lack of comprehensive data regarding the prevalence and distribution of procedural errors in endodontically treated teeth. This knowledge gap limits our understanding of how these errors differ between the maxilla and mandible and restricts the development of targeted strategies to enhance treatment quality and reduce failure rates.

Despite significant advancements in endodontic techniques and imaging modalities, procedural errors remain a critical challenge in achieving optimal treatment outcomes. These errors are particularly problematic in molar teeth due to their anatomical complexity and reduced accessibility. Although several international studies have evaluated the prevalence of endodontic procedural errors, there is limited research focusing specifically on the Egyptian subpopulation.

Understanding the patterns and frequencies of procedural errors in maxillary and mandibular teeth among Egyptians can aid clinicians in anticipating challenges, refining treatment strategies, and minimizing procedural failures. Moreover, differences in error distribution between the two jaws reported in other populations highlight the need for local investigation.

CBCT technology provides a detailed three-dimensional assessment of dental anatomy and procedural errors, offering superior diagnostic capabilities compared to two-dimensional radiography. This makes it an ideal tool for evaluating the prevalence and distribution of endodontic procedural errors.

Therefore, the aim of this study is to determine the prevalence and distribution of endodontic procedural errors in the maxilla and mandible using CBCT imaging in a selected Egyptian subpopulation.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans showing at least one permanent tooth that has undergone complete root canal treatment.
* Scans showing both jaw (maxilla and mandible) .
* Scans with good image quality and a voxel size of 0.2 mm or 0.3 mm.
* Egyptian nationals of either gender.
* Age over 18 years.

Exclusion Criteria:

* CBCT scans that do not show any teeth with complete root canal treatment.
* Completely edentulous patient.
* Low-quality images or scans with artefacts.
* Scans with voxel size larger than 0.3 mm.
* Non- Egyptian patients.
* Surgically treated endodontic cases (e.g., apicoectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of 379 CBCT scans obtained from Egyptian adult patients (over 18 years old) of both genders. These scans were acquired from radiology centers across Cairo, where patients were referred for various diagnostic purposes. The included scans represent cases with at least one fully endodontically treated permanent tooth and acceptable image quality
Sampling Method: Non-Probability Sample
Enrollment: 379 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Procedural Errors | Baseline assessment of all available cases within the study period
  Analysis of CBCT scans to detect and evaluate the prevalence of procedural errors such as instrument separation, perforations, ledges, and canal transportation in Endodontically treated teeth.

SECONDARY OUTCOMES:
Distribution of Procedural Errors between Maxilla and Mandible | Baseline assessment of all available cases within the study period.
  Analysis of CBCT scans to determine and compare the distribution of procedural errors, such as instrument separation, perforations, ledges, and canal transportation, between maxillary and mandibular teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Nehal N. Roshdy, Professor of Endodontics, Principal Investigator — Cairo University; Dr.sara, Lecturer in Endodontics, Study Chair — Cairo University

REFERENCES:
- [Background] Yousuf W, Khan M, Mehdi H. Endodontic Procedural Errors: Frequency, Type of Error, and the Most Frequently Treated Tooth. Int J Dent. 2015;2015:673914. doi: 10.1155/2015/673914. Epub 2015 Aug 10. PMID 26347779
- [Background] de Paula-Silva FW, Wu MK, Leonardo MR, da Silva LA, Wesselink PR. Accuracy of periapical radiography and cone-beam computed tomography scans in diagnosing apical periodontitis using histopathological findings as a gold standard. J Endod. 2009 Jul;35(7):1009-12. doi: 10.1016/j.joen.2009.04.006. PMID 19567324
- [Background] Patel S, Durack C, Abella F, Shemesh H, Roig M, Lemberg K. Cone beam computed tomography in Endodontics - a review. Int Endod J. 2015 Jan;48(1):3-15. doi: 10.1111/iej.12270. Epub 2014 Apr 2. PMID 24697513
- [Background] Nascimento EHL, Gaeta-Araujo H, Andrade MFS, Freitas DQ. Prevalence of technical errors and periapical lesions in a sample of endodontically treated teeth: a CBCT analysis. Clin Oral Investig. 2018 Sep;22(7):2495-2503. doi: 10.1007/s00784-018-2344-y. Epub 2018 Jan 21. PMID 29354883